CLINICAL TRIAL: NCT04143048
Title: A Study on Non-invasive Early Diagnosis of Gastrointestinal Stromal Tumors and Differentiation of Benign and Malignant Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-358
Record Dates: First submitted 2019-10-18; First posted 2019-10-29 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The construction of Gene detection technology flow: At this stage, a small panel targeted high-throughput sequencing process for gastrointestinal stromal tumors was established, and the association of tumor-associated mutation profiles in different patients with clinical stage was initially explored. It is planned to collect about 100 cases of gastrointestinal stromal tumors after surgery (freezing tissue or FFPE sections), DNA extraction and high-throughput sequencing of small panels, and analysis of the relationship between the mutation spectrum of each sample and the corresponding patient clinical data (staging).
  Interventions: Other: DNA extraction of tumer tissue samples and high-throughput sequencing of small panels
- Establishment of non-invasive gene testing technology process: In this stage, we plan to establish a small panel of peripheral blood cfDNA targeting high-throughput sequencing process, and verify the consistency of peripheral blood cfDNA and tissue gDNA in gene detection of gastrointestinal stromal tumors. About 50 patients were planned to be enrolled. Peripheral blood was collected once for each patient and the blood volume was 10mL. Meanwhile, the tumor tissue samples were collected within 5mm in diameter, depending on the size of the lesion . DNA extraction and small panel sequencing were performed for the two types of samples of the patients respectively, and the DNA sequencing results of the two types of samples were compared, and the clinical data of the corresponding patients were referenced to evaluate the consistency of the results of peripheral blood cfDNA and tissue gDNA for the gene detection of gastrointestinal stromal tumor.
  Interventions: Other: DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels
- Prospective cohort (double-blind recommended): Peripheral blood of about 150 patients was collected once and the blood volume was 10mL . Meanwhile, the tumor tissue samples were collected within 5mm in diameter, depending on the size of the lesion. Patients focus on the early stage of stromal tumors or those whose size under gastroenteroscopy is between 2 and 5 cm. DNA extraction and small panel sequencing were conducted for each patient sample. Based on the indicator results of the previous mutation spectrum for each stage of gastrointestinal stromal tumor, the clinical stage classification of patients and the benign and malignant nodules were determined by the mutation spectrum, and compared with the real clinical data of patients.
  Interventions: Other: DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels

INTERVENTIONS:
Other: DNA extraction of tumer tissue samples and high-throughput sequencing of small panels — DNA extraction of stromal tumor tissues and high-throughput sequencing of small panels were performed, and the relationship between the mutation spectrum of each sample and the corresponding patient clinical data (staging) was analyzed
  Groups: The construction of Gene detection technology flow
Other: DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels — DNA extraction and small panel sequencing were performed for the two types of samples of the patients respectively, and the DNA sequencing results of the two types of samples were compared, and the clinical data of the corresponding patients were referenced to evaluate the consistency of the results of peripheral blood cfDNA and tissue gDNA for the gene detection of gastrointestinal stromal tumor
  Groups: Establishment of non-invasive gene testing technology process
Other: DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels — DNA extraction and small panel sequencing were conducted for each patient sample. Based on the indicator results of the previous mutant spectrum for each stage of gastrointestinal stromal tumor, the clinical stage classification of patients and the benign and malignant nodules were determined by the mutant spectrum, and compared with the real clinical data of patients
  Groups: Prospective cohort (double-blind recommended)

SUMMARY:
Gastrointestinal Stromal Tumors (GIST) is the most common mesenchymal tumor of the gastrointestinal tract, and the incidence rate in China has increased year by year in recent years.Gastrointestinal stromal tumors are not sensitive to radiotherapy and traditional infusion chemotherapy. Currently, they are generally treated with surgery, but they are prone to recurrence and metastasis.For nodules with a particle size between 2 and 5 cm, there may be both benign and malignant, and there is still a lack of fast and accurate methods for distinguishing benign and malignant.Many benign nodules were removed (in the pathological examination of postoperative resected tissue). In addition, if it is found to be late, there is a possibility of invading surrounding tissues and metastasis, so that it is impossible to cure. Therefore, early diagnosis and early surgery and benign and malignant differentiation of small nodules are the key to the clinical diagnosis and treatment of gastrointestinal stromal tumors.At present, second-generation gene sequencing (NGS) and liquid biopsy are rarely reported in the field of GIST. A few domestic and foreign studies have found that it can detect rare mutation types, and may find secondary gene mutations early, which has potential applicability, but Overall, the clinical guidance of these NGS-based studies focuses on prognosis and drug resistance , as well as some studies based on low-throughput platforms. Therefore, early diagnosis and benign and malignant discrimination based on high-throughput sequencing and liquid biopsy have significant clinical significance for the diagnosis and treatment of gastrointestinal stromal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for stromal tumor resection
* Signed informed consent

Exclusion Criteria:

* the vital signs are not stable
* unconscious
* unwilling to cooperate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastrointestinal stromal tumor patients in Jiangsu Provincial People's Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Genetic mutations of patients with stromal tumor assessed by next-generation sequencing | 2019.8-2019.10
  DNA extraction of tumer tissue samples ,Preliminary exploration of tumor related mutation spectrum in different patients by gene sequencing

SECONDARY OUTCOMES:
Genetic mutations of patients with stromal tumor assessed by next-generation sequencing | 2019.11-2020.5
  DNA extraction of tumer tissue samples and blood tissue .To evaluate the consistency of peripheral blood cfDNA and tissue gDNA in gene detection of gastrointestinal stromal tumors,Using mutational spectra to determine the clinical stage of the patient and the benign and malignant small nodules

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China